CLINICAL TRIAL: NCT05946265
Title: Evaluation of Tooth Sensitivity After Scaling and Root Planing Treated With Photobiomodulation: a Randomized Controlled Double-blind Clinical Trial
Brief Title: Evaluation of Tooth Sensitivity After Scaling and Root Planing Treated With Photobiomodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Clinical Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: dental sensitivity
Record Dates: First submitted 2023-06-18; First posted 2023-07-14 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Photobiomodulation; Dental Hypersensitivity
Keywords: low-level light therapy; periodontal treatment
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Forty-four patients with dentin sensibility after non-surgical scaling and root planning (SRP) will be randomly included in 2 groups: Experimental Group: SRP+ Photobiomodulation (PBM) (660nm, 100W, area 0,5cm2, 200w/cm2, 30 seconds, 3 J, 6J/cm2. The primary outcome of the study will be the assessment of dentinal sensitivity after 7 days of RAR measured with the visual analog scale (VAS). The cutoff of VAS is 3. Also, it will be assessed the impact of oral health on the participant's quality of life, with the OHIP-14 questionnaire. The use of analgesics (paracetamol) will be prescribed as needed and the amount of medication will be calculated. These outcomes will be evaluated after 7 days and 1 month of application.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Immediately after periodontal treatment, the researcher responsible for applying the FBM will remove and open 1 envelope and perform the indicated procedure (FBM or simulation). Only this researcher will know the intervention applied to each patient. All other investigators will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention Group - RAR + FBM (n=56): The researcher responsible for FBM will remove the randomization envelope and apply Laser Therapy XP. All dosimetric parameters, details of sessions, and the number of FBM applications are presented in the project.
  Interventions: Device: Photobiomodulation
- Control Group (Placebo Comparator): Control Group - RAR + FBM simulation (n=56): Simulation of the use of FBM will be carried out identically to the Experimental group. The person responsible for applying the FBM will simulate irradiation by positioning the devices in the same locations described for the FBM group, however, the laser pointer will be turned off and the sound of the device will be recorded to mimic the use of the equipment and the participant will not identify the group to be used. who belongs. In this trial, we have no criteria for discontinuing or modifying allocated interventions because no harm is expected with this intervention. The study flowchart presents the details of the project
  Interventions: Device: simulation of Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — 120 patients with dentin sensibility after non-surgical scaling and root planning (SRP) will be randomly included in 2 groups: Experimental Group: SRP+ Photobiomodulation (PBM) The dosimetric parameters for the treatment included a wavelength of 660 nm applied in continuous mode with a radiant power of 100 mW (0.1 W). The irradiance ranged from 35.385 mW/cm² to 35 W/cm², with a beam area of 0.002826 cm². Each point received an exposure time of 30 seconds, resulting in a radiant exposure of 1.061 J/cm² and a total radiant energy of 3 J. The procedure involved six irradiated points per tooth, distributed across the vestibular surface (apical, middle, and cervical regions) and the palatal surface. The application technique was performed in contact, maintaining a 90-degree angle to the surface. The treatment consisted of a single session.
  Arms: Intervention group
Device: simulation of Photobiomodulation — Simulation of the use of FBM will be carried out identically to the Experimental group. The person responsible for applying the FBM will simulate irradiation by positioning the devices in the same locations described for the FBM group, however, the laser pointer will be turned off and the sound of the device will be recorded to mimic the use of the equipment and the participant will not identify the group to be used. who belongs. In this trial, we have no criteria for discontinuing or modifying allocated interventions because no harm is expected with this intervention.
  Arms: Control Group

SUMMARY:
One hundred twenty patients with dentin sensibility after non-surgical scaling and root planning (SRP) will be randomly included in 2 groups: Experimental Group: SRP+ Photobiomodulation (PBM) (660nm, 100W, area 0,5cm2, 200w/cm2, 30 seconds, 3 J, 6J/cm2. The study's primary outcome will be the assessment of dentinal sensitivity after 7 days of RAR measured with the visual analog scale (VAS). The cutoff of VAS is 3. The impact of oral health on the participant's quality of life will also be assessed with the OHIP-14 questionnaire. Analgesics (paracetamol) will be prescribed as needed, and the amount of medication will be calculated. These outcomes will be evaluated after 7 days and 1 month of application

DETAILED DESCRIPTION:
Objective: To evaluate tooth sensitivity after photobiomodulation in sensitive scaling and root planning treated teeth. Study design: Randomized, controlled, double-blind split-mouth clinical trial. Methods: One hundred twenty patients with dentin sensibility after non-surgical scaling and root planning (SRP) will be randomly included in 2 groups: Experimental Group: SRP+ Photobiomodulation (PBM). The dosimetric parameters for the treatment included a wavelength of 660 nm applied in continuous mode with a radiant power of 100 mW (0.1 W). The irradiance ranged from 35.385 mW/cm² to 35 W/cm², with a beam area of 0.002826 cm². Each point received an exposure time of 30 seconds, resulting in a radiant exposure of 1.061 J/cm² and a total radiant energy of 3 J. The procedure involved six irradiated points per tooth, distributed across the vestibular surface (apical, middle, and cervical regions) and the palatal surface. The application technique was performed in contact, maintaining a 90-degree angle to the surface. The treatment consisted of a single session.The primary outcome of the study will be the assessment of dentinal sensitivity after 7 days of RAR measured with the visual analog scale (VAS). The cutoff of VAS is 3. Also, it will be assessed the impact of oral health on the participant's quality of life, with the OHIP-14 questionnaire. The use of analgesics (paracetamol) will be prescribed as needed and the amount of medication will be calculated. These outcomes will be evaluated after 7 days and 1 month of application. If the data are normal, they will be submitted to the ANOVA test - one way. Data will be presented as means ± SD and the p-value will be set to < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 or older,
* diagnosed with periodontitis and experiencing dentin hypersensitivity greater than three on the VAS scale caused by a UNC-15 periodontal probe.
* both male and female patients were included,
* without comorbidities.

Exclusion Criteria:

* Patients taking medications that affect gingival metabolism (e.g., cyclosporine, phenytoin, nifedipine), inflammation (e.g., corticosteroids, anti-inflammatories), or pain (analgesics/NSAIDs),
* history of photosensitivity
* allergies to any medications used in the study.
* patients who experienced any complications during the study,
* allergic reactions to materials used or to paracetamol®
* Those who took any medication not provided in the study were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Pain (VAS) in baseline | baseline
  It will be evaluated through the application of the Visual Analog Scale (VAS) in which we will have a ruler with a length of 10 cm, without markings. One of the extremes is marked "0", and the other "100" which means respectively "no pain" and "unbearable pain".
  This ruler will be the same for all participants (a plasticized ruler where the patient marks with a permanent pen the amount of pain felt at that moment and this amount is measured in millimeters and the value noted in the patient's chart). Instructions on marking will always be given to the patient by the same operator. Each patient will be instructed to mark with a vertical line the point that best corresponds to the intensity of pain at the time of assessment . Without the presence of the patient, the operator will always measure with the same ruler, recording this data on the cards. This analysis will occur on all queries.
Pain (VAS) in 7 days | 7 days after treatment
  It will be evaluated through the application of the Visual Analog Scale (VAS) in which we will have a ruler with a length of 10 cm, without markings. One of the extremes is marked "0", and the other "100" which means respectively "no pain" and "unbearable pain".
  This ruler will be the same for all participants (a plasticized ruler where the patient marks with a permanent pen the amount of pain felt at that moment and this amount is measured in millimeters and the value noted in the patient's chart). Instructions on marking will always be given to the patient by the same operator. Each patient will be instructed to mark with a vertical line the point that best corresponds to the intensity of pain at the time of assessment . Without the presence of the patient, the operator will always measure with the same ruler, recording this data on the cards. This analysis will occur on all queries.
Pain (VAS) in 30 days | 30 days after treatment
  It will be evaluated through the application of the Visual Analog Scale (VAS) in which we will have a ruler with a length of 10 cm, without markings. One of the extremes is marked "0", and the other "100" which means respectively "no pain" and "unbearable pain".
  This ruler will be the same for all participants (a plasticized ruler where the patient marks with a permanent pen the amount of pain felt at that moment and this amount is measured in millimeters and the value noted in the patient's chart). Instructions on marking will always be given to the patient by the same operator. Each patient will be instructed to mark with a vertical line the point that best corresponds to the intensity of pain at the time of assessment . Without the presence of the patient, the operator will always measure with the same ruler, recording this data on the cards. This analysis will occur on all queries.

SECONDARY OUTCOMES:
Rescue medication at baseline | baseline
  Another parameter analyzed will be the number of analgesics ingested. At the beginning of the research, a pack of paracetamol® will be given to each participant , and use will be performed in case of pain. At the end of the experiment, the number of pills will be evaluated as another pain measurement parameter (drug tablet return). A procedure will be carried out to monitor the adherence of the participants (e.g., all patients will be asked to take the pack of analgesics to the consultation to check how they are being used).
Rescue medication at 7 days | 7 days after treatment
  Another parameter analyzed will be the number of analgesics ingested. At the beginning of the research, a pack of paracetamol® will be given to each participant , and use will be performed in case of pain. At the end of the experiment, the number of pills will be evaluated as another pain measurement parameter (drug tablet return). A procedure will be carried out to monitor the adherence of the participants (e.g., all patients will be asked to take the pack of analgesics to the consultation to check how they are being used).
Rescue medication at 30 days | 30 days after treatment
  Another parameter analyzed will be the number of analgesics ingested. At the beginning of the research, a pack of paracetamol® will be given to each participant , and use will be performed in case of pain. At the end of the experiment, the number of pills will be evaluated as another pain measurement parameter (drug tablet return). A procedure will be carried out to monitor the adherence of the participants (e.g., all patients will be asked to take the pack of analgesics to the consultation to check how they are being used).

CONTACTS AND LOCATIONS:
Overall Officials: Anna CR Horliana, PhD, Study Chair — University of Nove de Julho
Locations (1):
- Anna Carolina R.T. Horliana, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia Olazabal MV, Moya LEP, Cirisola RWC, Bruno LH, Safi FT, Ando-Suguimoto ES, Longo PL, Duran CCG, Bussadori SK, Motta LJ, Fernandes KPS, Mesquita-Ferrari RA, Horliana ACRT. Effect of photobiomodulation on dentin hypersensitivity: a randomized controlled double-blind clinical trial. Clin Oral Investig. 2025 Jan 24;29(1):84. doi: 10.1007/s00784-025-06149-z. PMID 39853488